CLINICAL TRIAL: NCT03341507
Title: A Comparative Study Between the Rigid Tube for Laryngoscopy, as a New Tool for Tracheal Intubation, and McIntosh Laryngoscope in Difficult Airway Patients
Brief Title: Tracheal Intubation With the Rigid Tube for Laryngoscopy- a New Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Marchis Ioan Florin, Principal Investigator, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIFlorin
Record Dates: First submitted 2017-11-03; First posted 2017-11-14 (Actual); Results first posted 2021-03-08 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-03

CONDITIONS: Intubation;Difficult
Keywords: laryngoscopy; retromolar
MeSH Terms: interventions — Laryngoscopy

STUDY DESIGN:
Intervention Model Description: A group of patients with difficult airway criteria will be intubated using the rigid tube for laryngoscopy. A classical laryngoscopy with a McIntosh laryngoscope will be performed prior intubation and the Cormack-Lehane grade of glottis visualisation will be noted. If the Cormack -Lehane grade of glotic visualisation 2b, 3 or 4, the intubation maneuvre is carried further with the rigid tube. If the Cormack-Lehane glottic visualisation grade is less than 2b (1 or 2a) the intubation is accomplished with the MacIntosh laryngoscope (conventional laryngoscope) and the patient is excluded from the study from that point further.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- laryngoscopy and tracheal intubation (Experimental): Tracheal intubation with the rigid tube for laryngoscopy for patients with difficult airway. Prior the use of rigid tube for laryngoscopy, a classical laryngoscopy with a McIntosh laryngoscope will be performed.
  Interventions: Device: classical laryngoscopy; Device: rigid tube for laryngoscopy

INTERVENTIONS:
Device: classical laryngoscopy — the laryngoscopy with the McIntosh laryngoscope performed prior the use of rigid tube and the Cormack-Lehane glottis visualisation noted.
  Other Names: laryngoscopy with McIntosh curved blade laryngoscope
Device: rigid tube for laryngoscopy — the view of glottis achieved with the rigid tub for laryngoscopy and tracheal intubation with an elastic gum bougie performed

SUMMARY:
This study evaluates the efficiency of the rigid tube for laryngoscopy for tracheal intubation in patients with presumed difficult airway and compare the classical laryngoscopy and this method in matter of glottis visualisation and tracheal intubation.

DETAILED DESCRIPTION:
The rigid tube for laryngoscopy is a 15 to 30 cm long metallic tube with a bevel end and a diameter of 0.5-2.0 cm , an instrument used to inspect the larynx and surrounding areas. It resembles a rigid bronchoscope but it is shorter. When in use, it has to be attached to a light source.

The hypothesis of the study stands that the rigid tube for laryngoscopy could be more efficient in tracheal intubation for difficult airway patients when the classical intubation with a curved blade laryngoscope is unsatisfactory.

The retromolar approach in both sides together with bougie(intubating tube introducer) intubation is the technique of intubation used in this study.

ELIGIBILITY:
Inclusion Criteria:

* patients with criteria of anatomically difficult airway from SARI (The Simplified Airway Risk Index Scale) parameters analysis
* patients with airway pathology which predicted difficult intubation: tumors or cervical masses, previous radiotherapy or surgery

Exclusion Criteria:

* stridor or marked laryngeal or tracheal stenosis, vocal cords polyps
* emergency surgery, decompensated cardiac or pulmonary disease
* grade 1 and 2a at classical laryngoscopy after Cormack- Lehane Classification

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ioan Florin Marchis, Md, Principal Investigator — University of Medicine and Pharmacy Iuliu Hatieganu- Cluj Napoca, Romania
Locations (1):
- Cluj County Emergency Hospital- ENT Clinic, Cluj-Napoca, Cluj, Romania

REFERENCES:
- [Background] Norskov AK, Rosenstock CV, Wetterslev J, Lundstrom LH. Incidence of unanticipated difficult airway using an objective airway score versus a standard clinical airway assessment: the DIFFICAIR trial - trial protocol for a cluster randomized clinical trial. Trials. 2013 Oct 23;14:347. doi: 10.1186/1745-6215-14-347. PMID 24152537
- [Background] Rutter JM, Murphy PG. Cormack and Lehane revisited. Anaesthesia. 1997 Sep;52(9):927. No abstract available. PMID 9349093

RESULTS

PARTICIPANT FLOW:
Groups:
- Laryngoscopy and Tracheal Intubation: Tracheal intubation with the rigid tube for laryngoscopy for patients with difficult airway. Prior the use of rigid tube for laryngoscopy, a classical laryngoscopy with a Mcintosh laryngoscope will be performed.
  classical laryngoscopy: the laryngoscopy with the Mcintosh laryngoscope performed prior the use of rigid tube and the Cormack-Lehane glottis visualisation noted.
  rigid tube for laryngoscopy: the view of glottis achieved with the rigid tub for laryngoscopy and tracheal intubation with an elastic gum bougie performed if the Cormack -Lehane glottis view is 2b,3 or 4 during conventional laryngoscopy
Period: Overall Study
Arm/Group | Laryngoscopy and Tracheal Intubation
Started | 64
Completed | 30
Not Completed | 34
Not completed — Cormack-Lehane grade 1 or 2a during conventional laryngoscopy | 34

BASELINE CHARACTERISTICS:
Population: Patients with difficult airway criteria according to SARI score schedulled for ear nose and throat (ENT) surgery under general anesthesia and tracheal intubation.
Groups:
- Tracheal Intubation With the Rigid Tube for Laryngoscopy: The study involved adult patients with ASA physical status 1-3, requiring surgery for an ENT pathology and having a presumed anatomically difficult airway according to The Simplified Airway Risk Index (SARI) score . Signed informed consent was obtained from all patients.
Arm/Group | Tracheal Intubation With the Rigid Tube for Laryngoscopy
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 64
  More than one race | 0
  Unknown or Not Reported | 0
The Simplified Airway Risk Index Scale(SARI) score ≥ 5. [Median (Inter-Quartile Range); unit: units on a scale] — The Simplified Airway Risk Index (or SARI) is a multivariate risk score for predicting difficult tracheal intubation. The SARI score ranges from 0 to 12 points, where a higher number of points indicates a more difficult airway. A SARI score of 4 or above indicate a difficult intubation. Seven parameters are used to calculate the SARI score: Mouth opening, thyromental distance, Mallampati score, movement of the neck, the ability to create an underbite, body weight and previous intubation history.
  units on a scale | 6 [5 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Time to Tracheal Intubation With the Rigid Tube
Description: the time from starting to use the rigid tube for laryngoscopy until the airway was secured.
Time Frame: 120 seconds
Population: Patients with a Cormack-Lehane grade 2b,3 or 4 during conventional laryngoscopy who had their airways secured with a rigid tube. Patients with a a Cormack-Lehane grade 1 and 2a were intubated with the curved blade laryngoscope and they were not included in analysis.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Laryngoscopy and Tracheal Intubation
Number analyzed (Participants) | 30
seconds | 50.5 [38 to 67]

2. Secondary Outcome: Complications During Intubation With Rigid Tube
Description: complications noticed during the use of rigid tube - hypoxia defined as oxygen saturation less than 80%
Time Frame: 5 minutes
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Laryngoscopy and Tracheal Intubation
Number analyzed (Participants) | 30
Participants | 1

3. Secondary Outcome: Late Complications of Intubation With Rigid Tube
Description: complications noticed following the use of rigid tube - sore throat, upper lip injury.
Time Frame: 3 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Laryngoscopy and Tracheal Intubation
Number analyzed (Participants) | 30
Participants | 8

4. Other Pre Specified Outcome: Conventional Laryngoscopy With the Curved Blade Laryngoscope ( MacIntosh) and Tracheal Intubation With the Curved Blade Laryngoscope if the Cormack-Lehane Glottis View Grade is 1 or 2a.
Description: Conventional laryngoscopy was performed with a MacIntosh curved blade laryngoscope, and the Cormack-Lehane grade of glottic visualization was registered. If the grade of glottis view according to Cormack-Lehane classification was less than 2b the patient was intubated using the curved blade laryngoscope. If the grade of glottic view was equal or more than 2b the tracheal intubation was carried further with the rigid tube.
Time Frame: 60 seconds
Population: Conventional laryngoscopy was performed with a MacIntosh curved blade laryngoscope, and the Cormack-Lehane grade of glottis visualization was registered. If the grade of glottis view according to Cormack-Lehane classification was less than 2b the patient was intubated using the curved blade laryngoscope. If the grade of glottis view was equal or more than 2b the tracheal intubation was carried further with the rigid tube.
Measure: Count of Participants; unit: Participants
Arm/Group | Laryngoscopy and Tracheal Intubation
Number analyzed (Participants) | 64
Participants | 34

ADVERSE EVENTS:
Time Frame: complications noticed during and following the use of rigid tube : time frame-3 days
Description: Complications during intervention- hypoxia, cardiac rhythm disturbances, hypertension, cardiac arrest, bronchospasm.
  Patient assessment after anesthesia for sore throat, voice disturbances, bleeding, teeth and soft tissue injury, neurological disorders following intervention, coughing, shortness of breath or chest pain
Arm/Group | Laryngoscopy and Tracheal Intubation
All-Cause Mortality (participants affected / at risk) | 0/64
Serious Adverse Events (participants affected / at risk) | 1/64
Other Adverse Events (participants affected / at risk) | 5/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laryngoscopy and Tracheal Intubation (N=64)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — hypoxia during airway management
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Laryngoscopy and Tracheal Intubation (N=64)
sore throat (Respiratory, thoracic and mediastinal disorders) | 5/30 (5) — complaint of sore throat after general anesthesia and tracheal intubation
upper lip injury (Skin and subcutaneous tissue disorders) | 3/30 (3) — upper lip small lesion after rigid tube intubation

LIMITATIONS AND CAVEATS:
This is an observational single-center study that relies on personal perception and the skill of a limited number of investigators. To master the rigid tube a period of training and regular use is needed.

The major disadvantage of the rigid tube for laryngoscopy is the reduced visual field which can be improved by increasing the tube diameter. The bougie intubation carries the risk of vocal cords injury and impossibility of advancing the tracheal tube if the respiratory space is too narrow.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT03341507/Prot_SAP_000.pdf